CLINICAL TRIAL: NCT00610064
Title: Brain Effects of Sacral Neuromodulation in Patients With Refractory Lower Urinary Tract Dysfunction
Brief Title: Brain Effects of Sacral Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Thomas M. Kessler, MD, Department of Urology, University of Bern, 3010 Bern
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KEK80_05; 1025
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Urinary Tract Disease
Keywords: Refractory lower urinary tract dysfunction; Sacral neuromodulation; Brain effects; Neuroimaging; Neuromodulation
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Baseline neuroimaging
  Interventions: Radiation: Baseline neuroimaging
- B (Other): Neuroimaging during sacral neuromodulation
  Interventions: Radiation: Neuroimaging during sacral neuromodulation

INTERVENTIONS:
Radiation: Baseline neuroimaging — Baseline neuroimaging using PET and MRI of the brain in patients before sacral neuromodulation
  Arms: A
Radiation: Neuroimaging during sacral neuromodulation — Neuroimaging during sacral neuromodulation using PET
  Arms: B

SUMMARY:
Sacral neuromodulation (SNM) has become an accepted treatment for patients with refractory lower urinary tract dysfunction such as urgency frequency syndrome, urgency incontinence, non-obstructive chronic urinary retention and chronic pelvic pain syndrome. Modulation of central afferent activity is considered critical to this therapeutic effect but the neural mechanisms are poorly understood.

We hypothesize that SNM has a significant effect on brain activity detectable by positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory lower urinary tract dysfunction scheduled for sacral neuromodulation

Exclusion Criteria:

* Pregnancy
* Age <18 years
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Effect of sacral neuromodulation on brain activity | 2-8 weeks

SECONDARY OUTCOMES:
Differences in brain activity effects of sacral neuromodulation (SNM) in patients with successful compared to failed SNM testing | immediately and 2-8 weeks after study inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Kessler, MD, Principal Investigator — Department of Urology, University of Bern, 3010 Switzerland
Locations (1):
- Department of Urology, University of Bern, Bern, Switzerland